CLINICAL TRIAL: NCT01173497
Title: A Phase II Study of the PARP Inhibitor, INIPARIB (BSI-201), in Combination With Chemotherapy to Treat Triple Negative Breast Cancer Brain Metastasis
Brief Title: A Study Evaluating INIPARIB in Combination With Chemotherapy to Treat Triple Negative Breast Cancer Brain Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11608; 20100210 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Estrogen Receptor Negative (ER-Negative) Breast Cancer; Progesterone Receptor Negative (PR-Negative) Breast Cancer; Human Epidermal Growth Factor Receptor 2 Negative (HER2-Negative) Breast Cancer; Brain Metastases
Keywords: Triple negative breast cancer; Brain metastasis; BSI-201; iniparib
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Triple Negative Breast Neoplasms | interventions — iniparib; Irinotecan

ARMS (1):
- INIPARIB, irinotecan (Experimental)
  Interventions: Drug: INIPARIB + irinotecan

INTERVENTIONS:
Drug: INIPARIB + irinotecan — 21 day cycle

SUMMARY:
The purpose of the study is to investigate the response rate for triple negative breast cancer patients with brain metastasis when INIPARIB is used in combination with irinotecan.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria -

1. Histologically-confirmed, ER negative, PR negative and Her2 negative adenocarcinoma of the breast with brain lesion on radiographic imaging.
2. ECOG Performance Status of 0-2.
3. Life expectancy of >12 weeks.
4. No limit to prior therapies with last anti-cancer treatment ≥ 2 weeks from initiation of protocol-based therapy provided all toxicities (other than alopecia) have resolved to ≤Grade 1 or baseline.
5. No active serious infection or other comorbid illness which would impair ability to participate in the trial.
6. Stable or decreasing dose of steroids for ≥ 7 days.
7. Interval ≥ 4 weeks between open brain biopsy and initiation of protocol-based therapy.
8. Patients must have adequate organ function.

Exclusion Criteria -

1. Pregnant or breast-feeding
2. Prior allergic reaction to INIPARIB
3. Prior allergic reaction to irinotecan.
4. Evidence of hemorrhage or impending herniation on baseline brain imaging
5. Evidence of diffuse leptomeningeal disease on brain MRI or by previously documented CSF cytology-NOTE: discrete dural metastases are permitted.
6. Clinically significant cardiac, renal, hepatic, infectious or pulmonary disease which might affect trial participation.
7. Concurrent or planned radiation, hormonal, chemotherapeutic, experimental or targeted biologic therapy.
8. Contraindication to gadolinium-enhanced MRI imaging.
9. Inability to comply with study and/or follow-up procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 months
  AS measured by intra or extra cranial time to progression (TTP)

SECONDARY OUTCOMES:
Response Rate | 12 months
  as measured by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (13):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - University of California At San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina-CH Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas